CLINICAL TRIAL: NCT05260983
Title: Preventing Type 2 Diabetes Through Using Acceptance and Commitment Therapy Principles to Target Illness Perceptions and Controllability Awareness in Educational Materials
Brief Title: Acceptance and Commitment Therapy Principles for Diabetes Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Principal Investigator, Megan Lipsett, Principal Investigator, University of Oregon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00000198
Record Dates: First submitted 2021-11-02; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: PreDiabetes; Diabetes Mellitus, Type 2; Diabetes; Diabetes type2
Keywords: diabetes; diabetes-related distress; diabetes self-management; illness perceptions; acceptance and commitment therapy; controllability awareness; psychological flexibility; body size stigma
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Prevention Education Only (Active Comparator): A brief standard diabetes prevention education engagement facilitation intervention modeled from the Center for Diseases Control and Prevention's National Diabetes Prevention Program.
  Interventions: Behavioral: Diabetes Prevention Education Only
- Diabetes Prevention Education and Acceptance and Commitment Therapy (Experimental): A brief diabetes prevention education and acceptance and commitment therapy engagement facilitation intervention. Acceptance and Commitment Therapy-informed materials (i.e. video, workbook, and activities) will retain facts about the condition, but will modify health messaging to clarify common inaccurate illness perceptions, reduce body size discrimination, and encourage psychological flexibility through framing illness perceptions, controllability awareness (i.e. ability to distinguish modifiable from unmodifiable components), non-judgmental awareness of what is occurring, willingness to allow experiences to occur, and the ability to step back from cognitions, acting according to personal values.
  Interventions: Behavioral: Diabetes Prevention Education and Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Diabetes Prevention Education and Acceptance and Commitment Therapy — A brief diabetes prevention education and acceptance and commitment therapy engagement facilitation intervention. Acceptance and Commitment Therapy-informed materials (i.e. video, workbook, and activities) will retain facts about the condition, but will modify health messaging to clarify common inaccurate illness perceptions, reduce body size discrimination, and encourage psychological flexibility through framing illness perceptions, controllability awareness (i.e. ability to distinguish modifiable from unmodifiable components), non-judgmental awareness of what is occurring, willingness to allow experiences to occur, and the ability to step back from cognitions, acting according to personal values.
  Arms: Diabetes Prevention Education and Acceptance and Commitment Therapy
Behavioral: Diabetes Prevention Education Only — A brief standard diabetes prevention education engagement facilitation intervention modeled from the Center for Disease Control and Preventions's National Diabetes Prevention Program.
  Arms: Diabetes Prevention Education Only

SUMMARY:
The investigators will evaluate whether a brief intervention (i.e. a workbook and video presenting educational information and activities materials for diabetes prevention) that incorporates principles drawn from focused Acceptance and Commitment Therapy frameworks impact positive and negative affect, stress perceptions, treatment expectations and intentions to engage, motivation and activation, illness perceptions, stress, diabetes distress, weight stigma internalization, controllability awareness, psychological flexibility, and self-efficacy - compared to standard diabetes prevention education materials.

DETAILED DESCRIPTION:
The investigators aim for this study to represent community-based, participatory research which is accessible, effective, understandable, and minimizing of stigma. Prior to conducting the study, the investigators will develop a community advisory board, consisting of practitioners who have expertise with the development and delivery of the intervention material and study population. Advisory board members will review the study materials and provide feedback for refining the study via meetings with the Principle Investigator. In addition, the investigators will hold a focus group composed of members of the community who have prediabetes or Type 2 Diabetes and who are interested in contributing to the study design. The focus group participants will review the study materials and provide feedback for improvement in understandability, minimizing stigma, effectiveness, access and relatability to the general public. Content from the community advisory board meetings and focus group will be used to inform the study design and will not be used for dissemination of data.

For the study implementation, the investigators will distribute online questionnaires on Amazon's Mechanical Turk and use CloudResearch service to recruit participants and manage the online project. Amazon's Mechanical Turk hosts research opportunities, called Human Intelligence Tasks, to online "workers". To distribute our surveys to this participant pool the investigators will embed our Qualtrics survey link in each Human Intelligence Tasks. The description of study purpose, time commitment, and research method will be available to the online "workers" who meet the inclusion criteria set on CloudResearch.

Participants will be assessed for eligibility (see below) via a qualtrics survey sent via Amazon Mechanical turk. As the eligibility process screens for risk of diabetes and assesses perceived stress, socioeconomic indicators, health status, and state anxiety, participants will also complete an initial consent form prior to eligibility screening. This process generates three distinct participant groups: study 1 ("Randomized Control Trial"), study 2 ("Cross-Sectional") and study 3 ("Sub-study"). The summary of measures given to each group is outlined in Table 1 below.

Study 1 ("Randomized Control Trial"): Participants will complete "pre-intervention measures" to assess individual differences (diabetes risk, diabetes program prevention participation, socioeconomic status, subjective social standing, co-morbidities, health status, illness perceptions, self-efficacy, and perceived stress). Participants will be randomized into either a brief standard diabetes education intervention or a brief diabetes education and acceptance and commitment therapy intervention. Acceptance and Commitment Therapy-informed materials will retain facts about the condition, but will modify health messaging (adapted from the Center for Diseases Control and Prevention's National Diabetes Prevention Program) to clarify common inaccurate illness perceptions, reduce body size discrimination, and encourage psychological flexibility through framing illness perceptions, controllability awareness (i.e. ability to distinguish modifiable from unmodifiable components), non-judgmental awareness of what is occurring, willingness to allow experiences to occur, and the ability to step back from cognitions, acting according to personal values. Following, participants will complete "post-intervention measures" to assess psychosocial variables (i.e. stress perceptions, treatment expectations and intentions to engage, motivation and activation, illness perceptions, acute stress, diabetes distress, diabetes locus of control, self-efficacy, controllability awareness, psychological flexibility, and self-efficacy).

ELIGIBILITY:
Inclusion Criteria:

1. United States Residency
2. 90% or higher Human Intelligence Task completion ratings (ratings which are assigned by mTurk researchers to workers upon completion of a Human Intelligence Task , and to indicate quality of worker history with mTurk).
3. At least 18 years of age
4. English-speaking
5. High-risk for Type 2 Diabetes, as indicated by a score of 5 or greater on the American Diabetes Association's diabetes risk test.

Exclusion Criteria:

1. Having been enrolled in a lifestyle program for diabetes prevention presently or within the past year.
2. Type 1 Diabetes diagnosis
3. Type 2 Diabetes diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
(Modified) Brief Diabetes Risk-Related Distress | Directly following the intervention
  The Diabetes Risk Distress Scale is a 5-item survey designed to measure patient concerns about diabetes prevention efforts and emotional burden of diabetes risk. The scale is modified for use in populations at high-risk of developing diabetes from the Brief Diabetes Distress Scale, with the inclusion of an additional item from the original 17-item Diabetes Distress Scale . Responses are collected using a 6-point likert scale ranging from "Not a problem" (1) to "A Very Serious Problem" (6), with higher scores reflecting higher levels of diabetes distress. Two subscales will also be considered: emotional burden and diabetes distress.
Brief Illness Perceptions Questionnaire | Directly following the intervention
  The Brief Illness Perceptions Questionnaire is a 9-item survey to rapidly assess the cognitive and emotional representations of illness tailored to focus on illness perceptions regarding diabetes risk. There are 5 items to measure cognitive representation of illness perceptions: consequences, timeline, personal control, treatment control, identity; two items to measure emotional representation: concern and emotional response; one item to measure illness comprehensibility / understanding; and one item designed to assess causal representation which asks participants to "rank-order the three most important factors that [the participant] believe caused [the participants] diabetes risk." Responses for the first 8 items are collected on an eleven-point Likert scale (e.g. Not at all affected emotionally (0) to Extremely affected emotionally (10)), where higher scores reflect a more extreme illness perception. Causal representation is an open-ended response.
Expected Diabetes Prevention-Related Controllability Awareness Scale | Directly following the intervention
  The Expected Diabetes Prevention-Related Controllability Awareness Scale is a 20- item survey designed to measure ''controllability awareness,": the extent to which the individual's behavioral and emotional responses to daily life situations reflect awareness of the controllable and uncontrollable aspects of the outcomes of those situations without focusing explicitly on controllability distinctions. The inventory was developed to assess controllability awareness as a characteristic of stress tolerance. The inventory consists of 20 simple statements assessing awareness of various aspects of controllability including personal control, shared control, others in control, and no one in control. Subjects indicate how much they agree or disagree with each statement from 1 = disagree strongly to 5 = agree strongly. Scores from all items are summed for a scoring running from 20-100, where higher scores reflect higher levels of controllability awareness.
Expected Program-Related Controllability Awareness Scale | Directly following the intervention
  The Expected Program-Related Controllability Awareness Scale was created to measure ''controllability awareness',": how much an individual's behavioral and emotional responses to daily life situations reflect awareness of the controllable and uncontrollable aspects of the outcomes of those situations without focusing explicitly on controllability distinctions. . Participants are provided a description of controllability awareness and then about the degree to which they agree with the statement "A diabetes prevention program like this one would help me prevent diabetes by teaching me to pay attention to the things about my situation that I can change and the things about my situation that I cannot change". Subjects indicate how much they agree or disagree with the statement on a 5-point scale from 1 = disagree strongly to 5 = agree strongly, where higher scores reflect higher controllability awareness.
Personalized Psychological Flexibility Index-Diabetes Prevention | Directly following the intervention
  The Personalized Psychological Flexibility Index-Diabetes Prevention is a 15-item survey designed to measure the ability to pursue valued life aims despite the presence of distress, which is a fundamental contributor to health. The index measures tendencies to avoid, accept, and harness discomfort during valued goal pursuit. For this study, we modified the scale to tailor the wording to goals related to diabetes prevention. In this study, three subscales are calculated: Avoidance subscale, Acceptance subscale, and Harnessing subscale. Items are measured on a 7 point likert scale of "strongly disagree" (1) to "strongly agree" (7). Psychological flexibility scores are computed by summing all items and range from 15-105, with higher scores reflecting more challenge in pursuing valued life goals despite presence of distress.
Brief Health Belief Model | Directly following the intervention
  The Brief Health Belief Model measure is designed to assess patient beliefs about the perceived seriousness ("If someone had Type 2 Diabetes or another related disease (such as stroke or heart disease), their whole life would change"), perceived susceptibility ("It is likely that I will get Type 2 Diabetes or another related disease (such as stroke or heart disease"), perceived prevention program benefits ("If I do a lifestyle change program for diabetes prevention it will decrease my chances of getting Type 2 Diabetes"), confidence ("I am confident that I could do what is recommended in the Diabetes Prevention Program if I wanted to"), and health motivation ("Maintaining good health is extremely important to me"). Each item is scored from 1 to 5 based on a Likert scale: "I strongly disagree" (1 point), "I disagree" (2 points), "I am not sure" (3 points), "I agree" (4 points), and "I strongly agree" (5 points).
Phenomenological Body Shame Scale - Revised | Directly following the intervention
  The Phenomenological Body Shame Scale - Revised is an 8 item survey derived from the original 18 item Phenomenological Body Shame Scale designed to measure the motivational and behavioral components of experiencing shame when participants imagine looking at themselves in a mirror, such as the desire to hide, escape, or disappear. Sample statements include "These diabetes education materials made me feel like covering my body." and "These diabetes education materials made me wish I were invisible." and are measured on a 5 point likert scale ranging from "not at all" scored as 1 to "extremely" scored as 5. Possible scores range from 8 to 40 with higher scores reflecting higher body shame.

SECONDARY OUTCOMES:
(Modified) 3-item Positive and Negative Affect | Directly following the intervention
  The Positive and Negative Affect Scale is a 20-item scale to assess momentary positive (e.g. active, excited, proud) and negative (e.g. afraid, scared, nervous) affect . We modified the Positive and Negative Affect Scale to be a brief 3-item version of the survey which measures overall positive and overall negative affect with examples reflecting the original scale items. This version additionally measures overall stress (e.g. out of control, overwhelmed by difficulties) during the intervention module. The items are prefaced with "While participating in this diabetes prevention module, to what extent did [the participant] feel:", followed by a likert scale ranging from very slightly or not at all (1) to extremely (5). Items for the brief 3-item Positive and Negative Affect Scale are considered individually and each score ranges from 1 to 5, with higher scores reflecting higher positive emotions, higher negative emotions, and higher stress.
Short-form State-Trait Anxiety Inventory | Directly following the intervention
  The Spielberger State-Trait Anxiety Inventory is a 6-item questionnaire designed and validated. It is a reliable and sensitive measure of anxiety. The 6-item version has been shown to have acceptable reliability , producing similar scores as the full 20-item inventory for those with normal and raised levels of anxiety. Participants are prompted to respond to indicate "how [the participant] feel right now, at this moment", followed by a list of common experiences (e.g. "I feel calm"," and "I am tense"). Responses range from Not at all (1) to Very much (4), with overall scores ranging from 20-80, where higher scores reflect higher states of anxiety.

OTHER OUTCOMES:
Treatment Expectations and Intentions to Engage | Directly following the intervention
  The teie survey is a 7-item survey that measures participant motivation, expectations, likelihood, confidence and perceived efficacy of a treatment program. Items were selected and adapted from previously validated measures designed to assess treatment expectancy and rationale credibility for use in clinical outcome studies. Credibility has been defined as 'how believable, convincing, and logical the treatment is, whereas expectancy refers to 'improvements that clients believe will be achieved" (Kazdin, 1979, as cited in Devilly & Borkovec, 2000). Participants see the following prompt: "The following questions ask about [the participants] feelings and intentions specifically after completing the previous activities." followed by a series of questions designed to assess confidence in the program, treatment credibility, intentions to engage, and perceived program efficacy. Responses are provided using a 5-point likert scale of Not at all(0) to Extremely(4).
Contemplation Ladder | Directly following the intervention
  The Contemplation Ladder is a single-item ladder to assess readiness to engage in lifestyle changes to prevent diabetes. The Contemplation Ladder is a visual analog composed of 11 rungs and 5 anchor statements, representing stages of change. For this study, the contemplation ladder anchor statements were altered to reflect stages of changes relevant to diabetes prevention behaviors. There are 10 rungs (with associated statements) that respondents use to indicate where they are along the stages of change. The response options correspond with the stage of precontemplation (e.g. "I have no thoughts about changing my health behaviors or enrolling in a prevention program."), contemplation, preparation, action, and maintenance (i.e. "I have changed my health behaviors and will never go back to the way I was before."). It is a brief measure of motivation or readiness to change, where (0) is the least motivated and (10) is the most motivated.
(Modified) Brief Patient Activation Measure | Directly following the intervention
  The (Modified) Brief Patient Activation Measure assesses patient self-reported knowledge for self-management of one's health or chronic condition, with a 22-item and a valid and reliable 13-item version . Belief in the importance of taking an active role ("When it comes to preventing diabetes, taking an active role in my own health care is the most important thing that affects my health"), has the confidence and knowledge to take action ("I know how to prevent diabetes."), has plans to take action ("I am confident that I will be able to maintain lifestyle changes to prevent diabetes, like healthy eating or exercising."), and has plans to stay the course under stress ("I am confident that I can maintain lifestyle changes, like healthy eating and exercising, even during times of stress."). Each item is rated on 4-point scale (1 strongly disagree to 4 strongly agree), where higher scores reflect higher levels of patient activation.
1-item Expected Diabetes Prevention Self-Efficacy Scale | Directly following the intervention
  The 1-item Expected Diabetes Prevention Self-Efficacy Scale was created for this study as a measure of self-efficacy related to expected diabetes prevention behaviors. This single item measure is intended to capture the extent that a person is able to control challenging environmental demands by taking adaptive action in diabetes prevention, following a brief engagement facilitation intervention. For this single item version, participants will be asked to respond about the degree to which they agree with the statement "When it comes to diabetes prevention, I am confident that I will be able to manage my diabetes risk to prevent Type 2 Diabetes (e.g. choose different foods and stick to a healthy eating pattern, keep my weight under control, get enough exercise, and visit my doctor once a year to monitor my diabetes risk)." with scores ranging from Not true at all (1) to Exactly true (4). Higher scores reflect higher perceived self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oregon - Social Affective Neuroscience Lab, Eugene, Oregon, United States

REFERENCES:
- [Derived] Lipsett M, Berkman E. A randomized controlled trial of an acceptance and commitment therapy-informed diabetes prevention program reduces body shame and distress. Health Psychol. 2025 May;44(5):549-559. doi: 10.1037/hea0001434. PMID 40232790